CLINICAL TRIAL: NCT01806571
Title: A Phase II Study of Combination Daunorubicin and Cytarabine (Ara-c) and Nilotinib (Tasigna) (DATA) in Patients Newly Diagnosed With Acute Myeloid Leukemia and KIT Overexpression
Brief Title: Daunorubicin Hydrochloride, Cytarabine, and Nilotinib in Treating Patients With Newly Diagnosed Acute Myeloid Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC1284; NCI-2013-00469 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 12-006178; MC1284 (Other: Mayo Clinic); P30CA015083 (NIH)
Record Dates: First submitted 2013-02-25; First posted 2013-03-07 (Estimated); Results first posted 2019-11-14 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Untreated Adult Acute Myeloid Leukemia
MeSH Terms: interventions — Cytarabine; Daunorubicin; nilotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (nilotinib, daunorubicin hydrochloride, cytarabine) (Experimental): INDUCTION THERAPY: Patients receive daunorubicin hydrochloride IV over 10 minutes on days 1-3, cytarabine IV continuously on days 1-7, and nilotinib PO BID on days 4-14. Patients achieving CR or CRi proceed to consolidation therapy. Patients not achieving a significant decrease in bone marrow recovery or CR/CRi upon bone marrow recovery receive another course of induction therapy.
  CONSOLIDATION THERAPY: Patients receive cytarabine IV every 12 hours on days 1, 3, and 5, and nilotinib PO BID on days 4-14. Treatment repeats every 28 days for 4 courses in the absence of disease progression or unacceptable toxicity. Patients achieving CR or CRi proceed to maintenance therapy.
  MAINTENANCE THERAPY: Patients receive nilotinib PO BID on days 1-84. Treatment repeats every 84 days for up to 8 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cytarabine; Drug: Daunorubicin Hydrochloride; Other: Laboratory Biomarker Analysis; Drug: Nilotinib; Other: Pharmacological Study

INTERVENTIONS:
Drug: Cytarabine — Given IV
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-Cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosar-U; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
Drug: Daunorubicin Hydrochloride — Given IV
  Other Names: Cerubidin; Cerubidine; Cloridrato de Daunorubicina; Daunoblastin; Daunoblastina; Daunoblastine; Daunomycin Hydrochloride; Daunomycin, hydrochloride; Daunorubicin.HCl; Daunorubicini Hydrochloridum; FI-6339; Ondena; RP-13057; Rubidomycin Hydrochloride; Rubilem
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Nilotinib — Given PO
  Other Names: AMN 107; Tasigna
Other: Pharmacological Study — Correlative studies

SUMMARY:
This phase II trial studies how well daunorubicin hydrochloride, cytarabine, and nilotinib work in treating patients newly diagnosed with acute myeloid leukemia. Drugs used in chemotherapy, such as daunorubicin hydrochloride and cytarabine, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Nilotinib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Giving daunorubicin hydrochloride with cytarabine and nilotinib may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the complete response rates of combination nilotinib, cytarabine, and daunorubicin (daunorubicin hydrochloride) in patients newly diagnosed with acute myeloid leukemia (AML) and v-kit Hardy-Zuckerman 4 feline sarcoma viral oncogene homolog (Kit) overexpression.

SECONDARY OBJECTIVES:

I. Determine the 2-year overall survival (OS) and disease-free survival (DFS) rates.

II. Determine the complete response duration in patients treated with this regimen.

III. Assess the safety and toxicity of this regimen based on National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.

TERTIARY OBJECTIVES:

I. Assess the prognostic and predictive factors (Kit mutation/expression level, fms-related tyrosine kinase 3 [Flt3] mutation) for patients treated with this regimen.

II. Assess the patterns of molecular response and relapse for Kit. III. Assess the effect on minimal residual disease (MRD) by polymerase chain reaction (PCR) or flow cytometry.

OUTLINE:

INDUCTION THERAPY: Patients receive daunorubicin hydrochloride intravenously (IV) over 10 minutes on days 1-3, cytarabine IV continuously on days 1-7, and nilotinib orally (PO) twice daily (BID) on days 4-14. Patients achieving complete remission (CR) or complete remission with incomplete blood count recovery (CRi) proceed to consolidation therapy. Patients not achieving a significant decrease in bone marrow recovery or CR/CRi upon bone marrow recovery receive another course of induction therapy.

CONSOLIDATION THERAPY: Patients receive cytarabine IV every 12 hours on days 1, 3, and 5, and nilotinib PO BID on days 4-14. Treatment repeats every 28 days for 4 courses in the absence of disease progression or unacceptable toxicity. Patients achieving CR or CRi proceed to maintenance therapy.

MAINTENANCE THERAPY: Patients receive nilotinib PO BID on days 1-84. Treatment repeats every 84 days for up to 8 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 6 months for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Untreated, histological confirmed acute myeloid leukemia (AML) based on World Health Organization (WHO) 2008 criteria with Kit expression (cluster of differentiation [CD] 117) of myeloblasts >= 20% by flow cytometry from bone marrow aspirate at diagnosis
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1, or 2
* Magnesium within normal limits (WNL)
* Potassium WNL
* Phosphorus WNL
* Serum amylase =< 1.5 x upper limit of normal (ULN)
* Serum lipase =< 1.5 x ULN
* Total bilirubin =< 1.5 x ULN (does not apply to patients with isolated hyperbilirubinemia [e.g., Gilbert's disease], in that case direct bilirubin should be =< 2 x ULN)
* Alkaline phosphatase =< 3 x ULN
* Serum glutamic-oxaloacetic transaminase (SGOT) (aspartate aminotransferase [AST]) =< 3 x ULN
* Creatinine =<1.5 x ULN
* Negative pregnancy test done =< 7 days prior to registration, for women of childbearing potential only
* Provide informed written consent
* Willing to return to consenting Mayo Clinic (Mayo Clinic's campus in Rochester, Mayo Clinic's campus in Arizona, or Mayo Clinic's campus in Florida) institution for follow-up during the active monitoring phase of the study
* Willing to provide bone marrow aspirate and blood samples for correlative research purposes

Exclusion Criteria:

* Any of the following because this study involves investigational agent(s) whose genotoxic, mutagenic and teratogenic effects on the developing fetus and newborn are unknown

  * Pregnant women
  * Nursing women
  * Men or women of childbearing potential who are unwilling to employ adequate contraception throughout the study and for 3 months after completion of study treatment
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Immunocompromised patients (other than that related to the use of corticosteroids) including patients known to be human immunodeficiency virus (HIV) positive
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, or psychiatric illness/social situations that would limit compliance with study requirements
* Receiving any other investigational agent which would be considered as a treatment for the primary neoplasm
* Other active malignancy =< 3 years prior to registration; EXCEPTIONS: non-melanotic skin cancer or carcinoma-in-situ of the cervix
* Previous treatment with chemotherapy or any other tyrosine kinase inhibitor for a hematological disorder; Exceptions: patients with prior diagnosis of myelodysplastic syndrome (MDS) and/or treatment with hypomethylating agent (azacytidine or decitabine) are not excluded, prior hydroxyurea allowed
* Impaired cardiac function including any one of the following:

  * Inability to monitor the QT interval on electrocardiogram (ECG)
  * Congenital long QT syndrome or a known family history of long QT syndrome
  * Clinically significant resting brachycardia (< 50 beats per minute)
  * Corrected QT (QTc) > 450 msec on baseline ECG; if QTc > 450 msec and electrolytes are not within normal ranges, electrolytes should be corrected and then the patient re-screened for QTc
  * Myocardial infarction =< 12 months prior to starting study
  * Other clinically significant uncontrolled heart disease (e.g. unstable angina, congestive heart failure or uncontrolled hypertension)
  * History of or presence of clinically significant ventricular, atrial tachyarrhythmias or ejection fraction cutoff
  * Left ventricle ejection fraction < 45%
  * History of, congestive heart failure requiring use of ongoing maintenance therapy for life-threatening ventricular arrhythmias
* Patients currently receiving treatment with strong cytochrome P450 family 3, subfamily A, polypeptide 4 (CYP3A4) inhibitors and treatment that cannot be either discontinued or switched to a different medication prior to starting study drug; patients receiving any medications or substances that are strong or moderate inhibitors of CYP3A4

  * Use of the following strong or moderate inhibitors is prohibited < 7 days prior to registration

    * Strong inhibitors of CYP3A4/5 > 5-fold increase in the plasma area under the curve (AUC) values or more than 80% decrease in clearance

      * Boceprevir (Victrelis)
      * Clarithromycin (Biaxin, Biaxin XL)
      * Conivaptan (Vaprisol)
      * Grapefruit juice
      * Indinavir (Crixivan)
      * Itraconazole (Sporanox)
      * Ketoconazole (Nizoral)
      * Lopinavir/ritonavir (Kaletra)
      * Mibefradil
      * Nefazodone (Serzone)
      * Nelfinavir (Viracept)
      * Posaconazole (Noxafil)
      * Ritonavir (Novir, Kaletra)
      * Saquinivir (Fortovase, Invirase)
      * Telaprevir (Incivek)
      * Telithromycin (Ketek)
      * Voriconazole (Vfend)
    * Moderate inhibitors of CYP3A4/5 > 2-fold in the plasma AUC values or 50-80% decrease in clearance

      * Amprenavir (Agenerase)
      * Aprepitant (Emend)
      * Atazanavir (Reyataz)
      * Ciprofloxacin (Cipro)
      * Darunavir (Prezista)
      * Diltiazem (Cardizem, Cardizem CD, Cardizem LA, Cardizem SR, Cartia XT, Dilacor XR, Diltia XT, Taztia XT, Tiazac)
      * Erythromycin (Erythrocin, E.E.S. , Ery-Tab, Eryc, EryPed, PCE)
      * Fluconazole (Diflucan)
      * Fosamprenavir (Lexiva)
      * Imatinib (Gleevec)
      * Verapamil (Calan, Calan SR, Covera-HS, Isoptin SR, Verelan, Verelan PM)
* Receiving any medications or substances that are inducers of CYP3A4; use of the following inducers are prohibited =< 7 days prior to registration

  * Strong inducers of CYP3A4/5 > 80% decrease in AUC

    * Avasimibe
    * Carbamazepine (Carbatrol, Epitol, Equetro, Tegretol, Tegretol-XR)
    * Phenytoin (Dilantin, Phenytek)
    * Rifampin (Rifadin)
    * St. John's wort
  * Moderate inducers of CYP3A4/5 50-80% decrease in AUC

    * Bosentan (Tracleer)
    * Efavirenz (Sustiva)
    * Etravirine (Intelence)
    * Modafinil (Provigil)
    * Nafcillin
    * Nevirapine (Viramune)
    * Phenobarbital (Luminal)
    * Rifabutin (Mycobutin)
    * Troglitazone
* Patients currently receiving treatment with any medications that have the potential to prolong the QT interval and the treatment cannot be either discontinued or switched to a different medication prior to starting study drug
* Impaired gastrointestinal (GI) function or GI disease that may significantly alter the absorption of study drug (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, small bowel resection or gastric bypass surgery)
* Acute or chronic pancreatic disease
* Known cytopathologically confirmed central nervous system (CNS) infiltration
* Acute or chronic liver disease or severe renal disease considered unrelated to the cancer
* History of significant congenital or acquired bleeding disorder unrelated to cancer
* Major surgery =< 4 weeks prior to registration of the study or who have not recovered from prior surgery
* Treatment with other investigational agents =< 14 days of registration
* Diagnosis of AML-M3 (or acute promyelocytic leukemia)

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2015-03-12 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2019-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aref Al-Kali, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic, Rochester, Minnesota

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Nilotinib, Daunorubicin Hydrochloride, Cytarabine): INDUCTION THERAPY: Patients receive daunorubicin hydrochloride IV over 10 minutes on days 1-3, cytarabine IV continuously on days 1-7, and nilotinib PO BID on days 4-14. Patients achieving CR or CRi proceed to consolidation therapy. Patients not achieving a significant decrease in bone marrow recovery or CR/CRi upon bone marrow recovery receive another course of induction therapy. CONSOLIDATION THERAPY: Patients receive cytarabine IV every 12 hours on days 1, 3, and 5, and nilotinib PO BID on days 4-14. Treatment repeats every 28 days for 4 courses in the absence of disease progression or unacceptable toxicity. Patients achieving CR or CRi proceed to maintenance therapy. MAINTENANCE THERAPY: Patients receive nilotinib PO BID on days 1-84. Treatment repeats every 84 days for up to 8 courses in the absence of disease progression or unacceptable toxicity. Cytarabine: Given IV Daunorubicin Hydrochloride: Given IV Laboratory Biomarker Analysis: Correlative studies Nilotinib: Given PO
Period: Overall Study
Arm/Group | Treatment (Nilotinib, Daunorubicin Hydrochloride, Cytarabine)
Started | 34
Completed | 34
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Nilotinib, Daunorubicin Hydrochloride, Cytarabine)
Number analyzed (Participants) | 34
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 58.6 [53 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 32
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Complete Responses (CR or CRi) During Induction Therapy
Description: The proportion of successes will be estimated by the number of successes divided by the total number of evaluable patients. Confidence intervals for the true success proportion will be calculated according to the approach of Duffy and Santner.
Time Frame: Up to 56 days
Measure: Number; unit: proportion of participants
Arm/Group | Treatment (Nilotinib, Daunorubicin Hydrochloride, Cytarabine)
Number analyzed (Participants) | 34
proportion of participants | 0.618

2. Secondary Outcome: Disease Free Survival(DFS) Rate
Description: Disease free survival time is defined for all evaluable patients who have achieved a CR or CRi as the time from registration to relapse or death due to any cause. The distribution of disease-free survival will be estimated using the method of Kaplan-Meier.
Time Frame: 35 months
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Treatment (Nilotinib, Daunorubicin Hydrochloride, Cytarabine)
Number analyzed (Participants) | 34
percentage of patients | 56.4 [41.6 to 76.6]

3. Secondary Outcome: Duration of Complete Response
Description: The distribution of duration of complete response will be estimated using the method of Kaplan-Meier.
Time Frame: 2 years
Population: Patients that acheived a complete response.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment (Nilotinib, Daunorubicin Hydrochloride, Cytarabine)
Number analyzed (Participants) | 21
Months | NA [30.4 to NA] — Median was not reached.

4. Secondary Outcome: Incidence of Adverse Events as Assessed by NCI CTCAE Version 4.0
Description: The maximum grade for each type of adverse event will be recorded for each patient, and frequency tables will be reviewed to determine patterns. Additionally, the relationship of the adverse event(s) to the study treatment will be taken into consideration. This data will be reported in the Adverse Events section of the results.
Time Frame: 35 months
Population: All treated patients
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Nilotinib, Daunorubicin Hydrochloride, Cytarabine)
Number analyzed (Participants) | 34
Participants | 34

5. Secondary Outcome: Overall Survival(OS) Rate
Description: Overall survival time is defined as the time from registration to death due to any cause. The distribution of survival time will be estimated using the method of Kaplan-Meier(Kaplan E 1958).
Time Frame: 39 Months
Measure: Number (95% Confidence Interval); unit: percentage of patients alive
Arm/Group | Treatment (Nilotinib, Daunorubicin Hydrochloride, Cytarabine)
Number analyzed (Participants) | 34
percentage of patients alive | 70.6 [55.7 to 87.3]

6. Other Pre Specified Outcome: Bone Marrow Flt3 Mutation
Description: Will be summarized and used to help characterize the types of patients accrued to this trial.
Time Frame: Baseline
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Bone Marrow Kit Mutation Status
Time Frame: Up to 3 years
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Bone Marrow Kit Mutation/Expression
Description: Will be summarized and used to help characterize the types of patients accrued to this trial.
Time Frame: Baseline
Reporting Status: Not Posted

9. Other Pre Specified Outcome: MRD, Assessed by PCR or Flow Cytometry
Description: MRD status will be correlated with response using Fisher's exact test. In addition, the relationship between MRD status (positive vs. negative) and disease-free survival will be evaluated using landmark analyses.
Time Frame: Up to 3 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were collected over 35 months and mortality was collected over 39 months.
Description: The descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 will be utilized for AE reporting.
Arm/Group | Treatment (Nilotinib, Daunorubicin Hydrochloride, Cytarabine)
All-Cause Mortality (participants affected / at risk) | 1/34
Serious Adverse Events (participants affected / at risk) | 31/34
Other Adverse Events (participants affected / at risk) | 34/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Nilotinib, Daunorubicin Hydrochloride, Cytarabine) (N=34)
Febrile neutropenia (Blood and lymphatic system disorders) | 18 (24)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Atrial flutter (Cardiac disorders) | 1 (1)
Heart failure (Cardiac disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 (1)
Jejunal hemorrhage (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Rectal fistula (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 1 (1)
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 1 (1)
Anorectal infection (Infections and infestations) | 2 (2)
Appendicitis (Infections and infestations) | 1 (1)
Catheter related infection (Infections and infestations) | 2 (2)
Enterocolitis infectious (Infections and infestations) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 3 (3)
Lung infection (Infections and infestations) | 4 (4)
Sepsis (Infections and infestations) | 5 (6)
Alanine aminotransferase increased (Investigations) | 7 (7)
Alkaline phosphatase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 5 (5)
Blood bilirubin increased (Investigations) | 5 (7)
Ejection fraction decreased (Investigations) | 1 (1)
Electrocardiogram QT corrected interval prolonged (Investigations) | 1 (1)
Lipase increased (Investigations) | 1 (1)
Serum amylase increased (Investigations) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (4)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 4 (5)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2)
Hypertension (Vascular disorders) | 5 (7)
Hypotension (Vascular disorders) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Nilotinib, Daunorubicin Hydrochloride, Cytarabine) (N=34)
Anemia (Blood and lymphatic system disorders) | 32 (72)
Febrile neutropenia (Blood and lymphatic system disorders) | 5 (5)
Cardiac disorders - Other, specify (Cardiac disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1)
Eye disorders - Other, specify (Eye disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 5 (7)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 3 (3)
Mucositis oral (Gastrointestinal disorders) | 5 (7)
Nausea (Gastrointestinal disorders) | 7 (7)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 4 (4)
Edema face (General disorders) | 1 (1)
Edema limbs (General disorders) | 2 (2)
Fatigue (General disorders) | 5 (6)
Fever (General disorders) | 3 (3)
Non-cardiac chest pain (General disorders) | 1 (1)
Catheter related infection (Infections and infestations) | 1 (1)
Lung infection (Infections and infestations) | 3 (4)
Skin infection (Infections and infestations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 15 (29)
Alkaline phosphatase increased (Investigations) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 15 (22)
Blood bilirubin increased (Investigations) | 20 (35)
CD4 lymphocytes decreased (Investigations) | 10 (23)
Creatinine increased (Investigations) | 1 (1)
Ejection fraction decreased (Investigations) | 1 (1)
Electrocardiogram QT corrected interval prolonged (Investigations) | 22 (36)
Lipase increased (Investigations) | 4 (4)
Lymphocyte count decreased (Investigations) | 15 (25)
Neutrophil count decreased (Investigations) | 34 (78)
Platelet count decreased (Investigations) | 34 (79)
Serum amylase increased (Investigations) | 1 (1)
Weight loss (Investigations) | 1 (1)
White blood cell decreased (Investigations) | 34 (77)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (4)
Hypocalcemia (Metabolism and nutrition disorders) | 3 (3)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 8 (8)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 3 (5)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1)
Scrotal pain (Reproductive system and breast disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 13 (20)
Purpura (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 25 (35)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertension (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-06): https://cdn.clinicaltrials.gov/large-docs/71/NCT01806571/Prot_SAP_000.pdf